CLINICAL TRIAL: NCT03966846
Title: The Effect of Regular Kefir Consumption on Metabolic Syndrome Parameters, Inflammatory Response, and Gut Microbiota: A Parallel-Group, Randomized, Controlled Clinical Study
Brief Title: Kefir and Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Hacettepe University (Other); Turkey Council of Higher Education Teaching Stuff Training Program (Unknown); Ege University (Other)
Responsible Party: Principal Investigator, Ezgi Bellikci Koyu, Assistant Professor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 152114
Record Dates: First submitted 2019-05-23; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Metabolic Syndrome; Obesity; Hypertension; Hyperlipidemias; Insulin Resistance
Keywords: probiotics; dairy products; kefir; gut microbiota
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Hypertension; Hyperlipidemias; Insulin Resistance | interventions — Kefir; Milk

STUDY DESIGN:
Intervention Model Description: There were two experimental groups. The kefir group, that received orally kefir, and the control group received milk
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kefir Group (Experimental): Kefir group received one bottle of kefir (180 ml) daily for 12 weeks. Microbial composition of the kefir included Lactococcus lactis ssp. lactis, Lactococcus lactis ssp. cremoris, Lactococcus lactis ssp. diacetylactis, Leuconostoc mesenteroides ssp. cremoris, Lactobacillus kefyr, Kliyveromyces marxianus, and Saccharomyces unisporus.
  Interventions: Dietary Supplement: Kefir
- Control Group (Placebo Comparator): Control group received one bottle of milk (180 ml) daily for 12 weeks.
  Interventions: Dietary Supplement: Milk

INTERVENTIONS:
Dietary Supplement: Kefir
  Arms: Kefir Group
Dietary Supplement: Milk
  Arms: Control Group

SUMMARY:
Metabolic syndrome is a cluster of metabolic disorders which increases the risk for diabetes and cardiovascular disease. In recent years, research has shown that probiotics may have positive effects on metabolic syndrome components. Although several health-promoting effects of kefir, have been suggested, there is limited evidence for its potential effect on metabolic syndrome. Therefore, it is necessary to clarify the effects of kefir on metabolic disorders including obesity, dyslipidemia, diabetes, and hypertension. To address the research gap, this study aimed to investigate the effects of daily kefir consumption on metabolic syndrome components, inflammatory response and gut microbiota composition in adults with MetS. The study was planned as a randomized, controlled, parallel design and completed with a total of 62 individuals who were diagnosed with metabolic syndrome according to the International Diabetes Federation (IDF) criteria. Participants were randomized into two groups and received daily 180 ml of kefir (n=31) or milk (as control) (n=31) for 12 weeks. Participants were assessed at baseline, week 4, week 8, and week 12 and at all controls dietary records, anthropometric measurements, and blood samples were collected. At baseline and 12th-week fecal samples were also collected in order to analyze gut microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old subjects
* Subjects diagnosed with metabolic syndrome according to the International Diabetes Federation (IDF) criteria.

Exclusion Criteria:

* Existence of lactose intolerance
* Existence of type 1 diabetes
* Existence of abnormal thyroid hormone levels
* Existence of chronic gastrointestinal system disease
* Existence of cancer
* Existence of severe liver disease
* Existence of kidney insufficiency
* Existence of immunodeficiency
* Taking medication to regulate blood glucose (except metformin) or lipid levels
* Taking antibiotics prior to one month of the study
* Consuming regular probiotic food or supplement
* Taking supplement which may affect the metabolic outcomes such as prebiotic or omega-3
* Dieting for weight loss or for another disease
* Being pregnant and breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Changes in lipid profile | baseline, week 4, week 8 and week 12
  Measurement of lipid profile (HDL cholesterol, triglyceride levels)
Changes in glycemic profile | baseline, week 4, week 8 and week 12
  Measurement of fasting glucose, insulin, and calculation of HOMA-IR
Changes in gut microbiota | week 0- week 12
  Determine the profile of gut flora (% abundance of various bacterial phyla, families, genera and species)

SECONDARY OUTCOMES:
Changes in Inflammatory Parametres | baseline and week 12
  Measurement of serum cytokines levels (high sensitive serum C- reactive protein ,TNF-α, IL-6, IL-10 ve IFN-γ)
Changes in serum cholesterol levels | baseline, week 4, week 8 and week 12
  Measurement of total cholesterol and its fractions (mg/dl)
Changes in triglycerides | baseline, week 4, week 8 and week 12
  Measurement of serum triglyceride (mg/dl)
Changes in lipoproteins | baseline and week 12
  Measurement of lipoproteins (mg/dl) (apolipoprotein A1, apolipoprotein B, lipoprotein (a))
Changes in homocysteine | baseline and week 12
  Measurement of homocysteine (umol/L)
Changes in glycated hemoglobin | baseline and week 12
  Measurement of HbA1c (%)
Changes in blood pressure | baseline, week 4, week 8 and week 12
  Measurement of systolic and diastolic blood pressure (mm Hg)
Changes in waist circumference | baseline, week 4, week 8 and week 12
  Measurement of waist circumference (cm)
Changes in Body Fat | baseline, week 4, week 8 and week 12
  Measurement of % body fat with BIA
Changes in BMI | baseline, week 4, week 8 and week 12
  weight and height will be measured to report BMI in kg/m2

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Bellikci-Koyu E, Sarer-Yurekli BP, Karagozlu C, Aydin-Kose F, Ozgen AG, Buyuktuncer Z. Probiotic kefir consumption improves serum apolipoprotein A1 levels in metabolic syndrome patients: a randomized controlled clinical trial. Nutr Res. 2022 Jun;102:59-70. doi: 10.1016/j.nutres.2022.02.006. Epub 2022 Mar 7. PMID 35405603